CLINICAL TRIAL: NCT06126939
Title: A Study on the Effect of Education Training on Parents With Autism Based on Denver Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Normal University (Other)
Responsible Party: Principal Investigator, lichao feng, Nurse practitioner, Hunan Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: lichaofeng
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Autism; Parents
Keywords: denver model; training; Intervention effect
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denver group (Experimental): In addition to routine health guidance, one-to-one parent classes were conducted to guide parents to interact with children once a week for 1h each time; A group leader was assigned to supervise the formulation of the intervention plan and ensure the quality of the intervention. The intervention lasted for 3 months
  Interventions: Behavioral: Educational training based on the Denver model
- Control group (No Intervention): Regular autism related knowledge health education

INTERVENTIONS:
Behavioral: Educational training based on the Denver model — In addition to routine health guidance, one-to-one parent classes were conducted to guide parents to interact with children once a week for 1h each time; A group leader was assigned to supervise the formulation of the intervention plan and ensure the quality of the intervention. The intervention lasted for 3 months
  Arms: Denver group

SUMMARY:
The goal of this clinical trial is to test the effects of parent training based on Denver model on parents' disease cognition level, coping style, parenting guilt, depression, anxiety and stress, quality of life, etc . The main question[s] it aims to answer are:

* What is the status quo of autistic parents' disease cognition level, coping style, parenting guilt, depression, anxiety and stress, and quality of life
* Whether education and training based on Denver model can improve autism parents' disease cognition level, coping style, parenting guilt, depression, anxiety and stress, and quality of life

Participants will receive educational training based on the Denver model. The researchers will compare the Denver model of early intervention with parents who receive regular autism health guidance to explore the effect of early intervention Denver model

ELIGIBILITY:
Inclusion Criteria:

* The child meets the diagnostic criteria for autism in the fifth edition of the American Diagnostic and Statistical Manual of Mental Disorders, and has been diagnosed by a physician；
* Parents of children aged 12-60 months with autism；
* Be the father or mother of the child, live with the child and take the main care of the child；
* Father ≥22 years old, mother ≥20 years old；
* Clear mind, normal intelligence, with normal cognitive ability.

Exclusion Criteria:

* Suffering from serious heart, liver and kidney diseases and mental illness;
* There are other family members suffering from serious illness or mental illness.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Trait Coping Style Questionnaire | One week before the intervention and one week after the intervention
  The questionnaire consists of 2 dimensions (positive coping and negative coping), with 10 entries in each dimension, using a 5-level rating (1 being definitely no, 5 being definitely yes). The higher the positive coping score, the more positive, and the higher the negative coping score, the more negative.
Illness Cognition Questionnaire-Parent version | One week before the intervention and one week after the intervention
  The scale includes three dimensions: helplessness, acceptance and perceived benefit, among which acceptance and perceived benefit belong to positive cognition, while helplessness belongs to negative cognition. Likert 1 to 4 scoring method was adopted for each item, and the 3 dimensions were scored respectively. The score range of each dimension was 6 to 24 points. The higher the score, the stronger the condition of the corresponding dimension, and the score of each dimension was not cumulative
Depression Anxiety Stress Scales | One week before the intervention and one week after the intervention
  There are 21 entries in total, 7 entries each for depression, anxiety and stress subscales. This scale is a 4-point Likert self-scoring scale, and the score of each question is between 0 and 3 points, "0" means "never", "1" means "sometimes", "2" means "often", and "3" means "always". The total score of each subscale multiplied by 2 is the final score. The higher the score, the more intense the negative emotional experience.
Guilt about Parenting Scale | One week before the intervention and one week after the intervention
  The scale is a single dimension scale with 10 items. All of them adopted the 7-point scoring method, and were assigned 1-7 points from completely non-conforming to completely conforming. The total score is 10 to 70, the higher the score, the higher the level of parenting guilt of the subject
Beach Center Family Quality of Life Scale | One week before the intervention and one week after the intervention
  The scale included 25 items in 5 dimensions, including family interaction (6 items), parenting (6 items), emotional health (4 items), physical/material welfare (5 items) and support related to disability (4 items). Likert5-level scores were used, from "very dissatisfied" to "very satisfied", 1-5 points were assigned, with a total score of 25 to 125 points. The higher the score, the more satisfied the individual was with the quality of family life.

IPD SHARING:
Plan to Share IPD: Undecided